CLINICAL TRIAL: NCT02300480
Title: Effects of Calot's Triangle Block for Postoperative Analgesia in Patients Undergoing Laparoscopic Cholecystectomy: a Prospective, Randomized, Double-blind, Controlled, Clinical Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Min Su, The Department of Anesthesiology and Pain Medicine, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CYYYMZ-005
Record Dates: First submitted 2014-11-19; First posted 2014-11-25 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Post-operative Pain; Gallstone Disease
Keywords: pain; calot's triangle; local block; analgesia; patient controlled intravenous analgesia
MeSH Terms: conditions — Pain, Postoperative; Cholelithiasis; Pain; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTB group (Experimental): Participants in this group will receive a single injection for calot's triangle block combined with PCIA post-operatively. CTB will be conducted by bile duct needle and 1.0% 10 ml ropivacaine will be injection in calot's triangle when before surgical dissection.Participants in this group will also receive PCIA after surgery,the regimens of PCIA are included tramadol 800 mg, flurbiprofenaxetil 100 mg with normal saline added up to a volume of 80 ml in total.
  Interventions: Procedure: CTB group
- PCIA group (Active Comparator): Participants in this group will receive PCIA post-operatively (tramadol 800 mg and flurbiprofen axetil 100mg with normal saline added up to a volume of 80ml in total ) .The PCIA pump was set up with a 5 ml loading dose, a 2 ml bolus dose, a 15 min lockout interval and background infusion at a rate of 1 ml/h.
  Interventions: Procedure: PCIA group

INTERVENTIONS:
Procedure: CTB group — CTB: A single injection of 1.0% 10ml ropivacaine by bile duct needle in calot's triangle when before surgical dissection.After surgery,participants in this group will also receive PCIA.
  Arms: CTB group
Procedure: PCIA group — The formula of the PCIA included tramadol 800 mg, flurbiprofen axetil 100mg with saline added up to a volume of 80 ml in total. The PCIA pump was set up with a 5 ml loading dose, a 2 ml bolus dose, a 15 min lockout interval and background infusion at a rate of 1 ml/h.
  Arms: PCIA group

SUMMARY:
Chronic pain after laparoscopic cholecystectomy (LC) is a common complication with an incidence ranging between 3-56%. In many cases, however, the cause chronic pain after LC remains unknown and visceral hyperalgesia and central sensitization have been suggested to be part of the pathophysiology. So the purpose of this study is to determine whether Calot's Triangle Block (CTB) combined with patient controlled intravenous analgesia (PCIA) is superior to PCIA in reducing the incidence of chronic pain after LC.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is currently regarded as the gold standard treatment for symptomatic gallstone disease. Compared with open cholecystectomy, LC benefits include less postoperative pain, reduced analgesic consumption, and earlier discharge. However, besides the advantages mentioned above, there are exist complexity and diversity of the acute pain after LC, which consists of a somatic, a visceral and a referred pain component. Meanwhile, our team also found many LC patients experience visceral pain after surgery. According to epidemic research show that chronic pain after LC is a common complication with an incidence ranging between 3-56%. Several reports have indicated that early postoperative pain has been shown to be a significant risk factor of chronic pain. In many cases, however, the cause chronic pain after LC remains unknown and visceral hyperalgesia and central sensitizationhave been suggested to be part of the pathophysiology. To reduce the incidence of chronic pain after LC, so we conduct the randomized controlled trial to investigate whether calot's triangle block combined with PCIA is superior to PCIA in reducing the incidence of chronic pain after LC.

This study was approved by the institutional review board of the First Affiliated Hospital of Chongqing Medical University. The protocol design is in accordance with Consolidated Standards of Reporting Trials (CONSORT) statement. All potentially eligible participants will be asked to give written informed consent before they are enrolled in this study. This study is a prospective, randomized, double-blind, controlled clinical trial guided by the standard of good clinical practice (GCP), and eligible participants are divided into two groups: group CTB and group PCIA, and primary assess the outcomes of the incidence of chronic pain after LC and the intensity of acute pain after LC.

Participants in group CTB will receive a single injection of ropivacaine in calot's triangle before surgical dissection combined with PCIA post-operatively.

Participants in group PCIA will receive a single injection in calot's triangle with normal saline before surgical dissection and PCIA post-operatively.

The primary outcome of this study is the incidence of chronic pain after LC.

The secondary outcomes of this study are acute post-operative pain, moderate-severe pain, rescue medication and adverse events associated with the post-operative analgesia.

This study will be conducted under the supervision of an independent auditor. Every week, the auditor checked the data of the participants the day after the surgery was conducted. Assessment of pain intensity and prognostic outcomes must be confirmed by the auditor in sample population. When there is disagreement between surgeon and anesthesiologists in evaluating the prognosis of patients, the auditor must solve this disagreement by discussion with evaluators. Data will be double-entered by two statisticians with limitation of access and locked during statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* men or woman over 18 the years and younger than 65 years old who will receive selective laparoscopic cholecystectomy.

Exclusion Criteria:

* age below 18 years or over 65 years
* American Society of Anesthesiologists grade III or greater
* Diabetes
* chronic pain of any kind other than gallbladder disease
* allergic to local anesthetics
* cognitive impairment or communication problems
* peptic ulcer
* received opioids、NSAID or tranquilizers (treatment for over 1 wk before the cholecystectomy)
* history of alcohol or drug abuse
* the operation was converted to an open procedure
* gangrenous cholecystitis
* common bile duct exploration or insertion of a T-drain
* other invasive procedures
* severe hepatic or renal impairment
* post-operative severe complications(e.g. pyogenic infection)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-08 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Chronic post-surgical pain | 3 months post-operatively
  Chronic post-surgical pain intensity will be measured as more than 3 months by numerical rating scale (NRS) for pain

SECONDARY OUTCOMES:
Acute pain post-operatively | 2h,4h,6h,12h,24h, 48h post-operatively
  Pain intensity will be measured by visual analogue scale(VAS)
Analgesic Rescue | from 2h to 48h post-operatively
  The dosages of opioid or non-opioid analgesic rescue medications
Adverse events associated with post-operative analgesia | from 2h to 48h post-operatively
  incomplete analgesia; nausea and vomiting; respiratory depression; over-sedation
moderate-severe pain | 3,6months postoperatively
  Pain intensity will be measured by numerical rating scale (NRS)
chronic post-surgical pain | 6months postoperatively
  chronic post-surgical pain intensity will be measured by numerical rating scale (NRS) for pain

CONTACTS AND LOCATIONS:
Overall Officials: Su Min, MD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- China,Chongqing The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Background] Blichfeldt-Eckhardt MR, Ording H, Andersen C, Licht PB, Toft P. Early visceral pain predicts chronic pain after laparoscopic cholecystectomy. Pain. 2014 Nov;155(11):2400-7. doi: 10.1016/j.pain.2014.09.019. Epub 2014 Sep 22. PMID 25250720
- [Background] Bisgaard T, Klarskov B, Rosenberg J, Kehlet H. Characteristics and prediction of early pain after laparoscopic cholecystectomy. Pain. 2001 Feb 15;90(3):261-269. doi: 10.1016/S0304-3959(00)00406-1. PMID 11207398
- [Background] Lamberts MP, Lugtenberg M, Rovers MM, Roukema AJ, Drenth JP, Westert GP, van Laarhoven CJ. Persistent and de novo symptoms after cholecystectomy: a systematic review of cholecystectomy effectiveness. Surg Endosc. 2013 Mar;27(3):709-18. doi: 10.1007/s00464-012-2516-9. Epub 2012 Oct 6. PMID 23052498
- [Background] Macrae WA. Chronic pain after surgery. Br J Anaesth. 2001 Jul;87(1):88-98. doi: 10.1093/bja/87.1.88. No abstract available. PMID 11460816
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Joris J, Thiry E, Paris P, Weerts J, Lamy M. Pain after laparoscopic cholecystectomy: characteristics and effect of intraperitoneal bupivacaine. Anesth Analg. 1995 Aug;81(2):379-84. doi: 10.1097/00000539-199508000-00029. PMID 7618731
- [Background] Bisgaard T, Rosenberg J, Kehlet H. From acute to chronic pain after laparoscopic cholecystectomy: a prospective follow-up analysis. Scand J Gastroenterol. 2005 Nov;40(11):1358-64. doi: 10.1080/00365520510023675. PMID 16334446
- [Background] Ingelmo PM, Bucciero M, Somaini M, Sahillioglu E, Garbagnati A, Charton A, Rossini V, Sacchi V, Scardilli M, Lometti A, Joshi GP, Fumagalli R, Diemunsch P. Intraperitoneal nebulization of ropivacaine for pain control after laparoscopic cholecystectomy: a double-blind, randomized, placebo-controlled trial. Br J Anaesth. 2013 May;110(5):800-6. doi: 10.1093/bja/aes495. Epub 2013 Jan 4. PMID 23293276
- [Background] Donatsky AM, Bjerrum F, Gogenur I. Intraperitoneal instillation of saline and local anesthesia for prevention of shoulder pain after laparoscopic cholecystectomy: a systematic review. Surg Endosc. 2013 Jul;27(7):2283-92. doi: 10.1007/s00464-012-2760-z. Epub 2013 Jan 26. PMID 23355159
- [Background] Gurusamy KS, Nagendran M, Guerrini GP, Toon CD, Zinnuroglu M, Davidson BR. Intraperitoneal local anaesthetic instillation versus no intraperitoneal local anaesthetic instillation for laparoscopic cholecystectomy. Cochrane Database Syst Rev. 2014 Mar 13;(3):CD007337. doi: 10.1002/14651858.CD007337.pub3. PMID 24627292
- [Background] Desautels SG, Slivka A, Hutson WR, Chun A, Mitrani C, DiLorenzo C, Wald A. Postcholecystectomy pain syndrome: pathophysiology of abdominal pain in sphincter of Oddi type III. Gastroenterology. 1999 Apr;116(4):900-5. doi: 10.1016/s0016-5085(99)70073-9. PMID 10092312
- [Background] Woolf CJ. Central sensitization: implications for the diagnosis and treatment of pain. Pain. 2011 Mar;152(3 Suppl):S2-S15. doi: 10.1016/j.pain.2010.09.030. Epub 2010 Oct 18. PMID 20961685
- [Background] Shaffer E. Acalculous biliary pain: new concepts for an old entity. Dig Liver Dis. 2003 Jul;35 Suppl 3:S20-5. doi: 10.1016/s1590-8658(03)00089-6. PMID 12974505
- [Background] SHAFIROFF BG, HINTON JW. Surgical anatomy of the choledochal nerves. Arch Surg (1920). 1950 May;60(5):944-952. doi: 10.1001/archsurg.1950.01250010967009. No abstract available. PMID 15411317
- [Background] Womack NA, Crider RL. The Persistence of Symptoms Following Cholecystectomy. Ann Surg. 1947 Jul;126(1):31-55. doi: 10.1097/00000658-194707000-00004. No abstract available. PMID 17858976
- [Background] Kellow JE. Sphincter of Oddi dysfunction type III: another manifestation of visceral hyperalgesia? Gastroenterology. 1999 Apr;116(4):996-1000. doi: 10.1016/s0016-5085(99)70086-7. No abstract available. PMID 10092325
- [Background] Kurucsai G, Joo I, Fejes R, Szekely A, Szekely I, Tihanyi Z, Altorjay A, Funch-Jensen P, Varkonyi T, Madacsy L. Somatosensory hypersensitivity in the referred pain area in patients with chronic biliary pain and a sphincter of Oddi dysfunction: new aspects of an almost forgotten pathogenetic mechanism. Am J Gastroenterol. 2008 Nov;103(11):2717-25. doi: 10.1111/j.1572-0241.2008.02068.x. Epub 2008 Aug 5. PMID 18684173
- [Background] Hickey OT, Burke SM, Hafeez P, Mudrakouski AL, Hayes ID, Shorten GD. Severity of acute pain after breast surgery is associated with the likelihood of subsequently developing persistent pain. Clin J Pain. 2010 Sep;26(7):556-60. doi: 10.1097/AJP.0b013e3181dee988. PMID 20639740
- [Background] Katz J, Jackson M, Kavanagh BP, Sandler AN. Acute pain after thoracic surgery predicts long-term post-thoracotomy pain. Clin J Pain. 1996 Mar;12(1):50-5. doi: 10.1097/00002508-199603000-00009. PMID 8722735